CLINICAL TRIAL: NCT04748796
Title: Comparison of Landiolol Versus Standard of Care for Prevention of Mortality in Patients Hospitalized for a Septic Shock With Hypercontractility: an Open Label Prospective Randomized Study
Brief Title: Comparison of Landiolol Versus Standard of Care for Prevention of Mortality in Patients Hospitalized for a Septic Shock With Hypercontractility
Acronym: HyperBetashock
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: CH Dieppe (Unknown); CH Elbeuf (Unknown); CH Le Havre (Unknown); Centre Hospitalier de Beauvais (Other); CH Compiègne (Unknown); CH Laon (Unknown); University Hospital, Caen (Other); CH Cherbourg (Unknown); University Hospital, Lille (Other); CH Douai (Unknown); CH Montreuil (Unknown); Centre Hospitalier de Roubaix (Other); Centre Hospitalier de Bethune (Network); CH Lomme (Unknown); Centre Hospitalier de Lens (Other); Tourcoing Hospital (Other); Centre Hospitalier VALENCIENNES (Other); Centre Hospitalier Arras (Other); Hospital Ambroise Paré Paris (Other); University Hospital, Brest (Other); Henri Mondor University Hospital (Other); Hospital Avicenne (Other); University Hospital, Montpellier (Other); CH Calais (Unknown); Hôpital Edouard Herriot (Other); Centre Hospitalier Universitaire de Nīmes (Other); Groupe Hospitalier Pitié-Salpêtrière (Unknown); Hôpital Louis Mourier, Colombes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2020_843_0057
Record Dates: First submitted 2021-01-27; First posted 2021-02-10 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Septic Shock; Tachycardia; Mortality During Septic Shock; Beta-blocker
Keywords: Septic Shock; Tachycardia; mortality during septic shock; beta-blocker
MeSH Terms: conditions — Shock, Septic; Tachycardia | interventions — landiolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 2 days with landiolol IV + usual care
  Interventions: Drug: Landiolol
- Control group (Active Comparator): usual care according to the attending physician and following the guidelines of surviving sepsis campaign.
  Interventions: Other: echocardiography

INTERVENTIONS:
Other: echocardiography — Full echocardiography will be performed at baseline and during the follow-up at H1, H3, H6 and H12.
  Arms: Control group
Drug: Landiolol — Patients randomized to the experimental group will be treated according to the standard of care plus for 2 days with landiolol IV started at a dose of 1 microgram/kg/min and progressively increased every 10 minutes to a maximum of 40 micrograms/kg/min.
  Arms: Experimental group

SUMMARY:
Several data emphasize the relation between tachycardia (>90/min) and high mortality during septic shock. The investigators previously demonstrated the high mortality associated with hypercontractility, tachycardia and the presence of a left ventricular obstruction. A severe hypovolemia, a hyper adrenergic stimulation or a severe vasoplegia can all explain this relation between tachycardia, hypercontractility and the mortality during septic shock.

Landiolol is another short-term acting beta-blocker with a half-life of 4 minutes without any beta 2 activity or membrane stabilizing effect. The landiolol has been used in critically ill patients to control supraventricular tachycardia but not in this context of tachycardia and septic shock. The investigators hypothesize that landiolol by reducing the heart rate may improve the survival of patients treated for a septic shock and presenting with an hypercontractility state.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient admitted for a septic shock (according to the SEPSIS3 definition: sepsis with persisting hypotension (MAP<65mmHg or SAP <90mmHg) requiring vasopressors to maintain MAP>65mmHg and having a serum lactate level >2 mmol/L
* Patient who received at least 30ml/kg of fluid and absence of fluid responsiveness
* Left ventricular ejection fraction >65% (visual or Simpson method using echocardiography)
* Tachycardia >100 bpm in sinus rhythm with a MAP 65mmHg for more than 1 hour
* Patient receiving invasive mechanical ventilation
* Patients adapted to the ventilator under sedation and analgesia
* Written informed consent
* Patient covered by French national health insurance

Exclusion Criteria:

* Patients with inclusion criteria already present for more than 36 hours
* Patient treated with Dobutamine, adrenaline or isoprenaline
* Patient currently treated with beta blockers (previous home betablocker treatment is not an exclusion criteria)
* Supra ventricular (atrial fibrillation or flutter) or ventricular arrhythmias
* Patients with any form of cardiac pacing
* Sick sinus syndrome
* Severe atrioventricular (AV) nodal conductance disorders (without pacemaker): 2nd or 3rd degree AV block
* Known pulmonary hypertension
* ScVO2 <70%
* Moribund
* Cardiac arrest
* Non-treated phaeochromocytoma
* Acute asthmatic attack
* Pregnant or breastfeeding woman
* Patient deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision),
* Age <18 years
* Hypersensitivity to the active substance or to any of the excipients
* Severe bradycardia (less than 50 beats per minute)
* Cardiogenic shock
* Severe hypotension
* Decompensated heart failure when considered not related to the arrhythmia
* Severe, uncorrectable metabolic acidosis
* Presence of significant bleeding, or
* Acute respiratory distress defined by increased oxygen dependency, polypnea > 30 /min, signs of struggle (pulling, thoraco-abdominal sway) if the patient is not intubated and ventilated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Variation of mortality rate in landiolol group compared to control group | day 28

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No